CLINICAL TRIAL: NCT05778136
Title: Exercise in Lung Cancer Patients - Specific Training, Muscle Mass and Force Development
Brief Title: Lung Cancer, Exercise and Force Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Quist, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MQCLFW; H-22073691 (Other: The Scientific Ethics Committee)
Record Dates: First submitted 2023-03-01; First posted 2023-03-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: Exercise; Functionality; Resistance training; Muscle, skeletal; Sarcopenia
MeSH Terms: conditions — Lung Neoplasms; Motor Activity; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel assignment. The participants will be randomized to either left or right leg resistance training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants receive usual care
- Usual Care + exercise (Experimental): Participants receive usual care and one-leg resistance exercise training
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Supervised resistance training. 2 sessions/week for 12 weeks. The exercises are one-legged leg-press and one-leg knee extension. Resistance training start-up phase comprises 3 sets of 10 repetitions in each of the two exercises with 50% of 1RM. Resistance training progressive phase comprises 3 sets (leg-press) of 5-8 repetitions (70-90% 1 RM) and 6 sets (knee extension) of 8 repetition (75% 1RM). Rest between sets: 3 minutes
  Arms: Usual Care + exercise

SUMMARY:
This study evaluates the effectiveness of a supervised one-leg resistance training program in patients with inoperable lung cancer with the primary outcome being rate of force development.

Study design: Single center, two-armed, parallel-group, randomized controlled trial. The primary outcome being rate of force development after 12 weeks of progressive resistance training.

DETAILED DESCRIPTION:
Muscular dysfunction and sarcopenia are known phenomena in cancer patients, and patients experience reduced muscle function and muscle loss regardless of cancer type or stage. Studies indicate that there are a number of cancer-specific and non-cancer-specific factors that influence muscle dysfunction, such as age, poor nutrition, physical inactivity, cancer pathology and treatment preparations. The decreased muscle function can ultimately lead to cachexia, typically seen in stage III - IV lung cancer patients.

Previous studies have focused on 1-RM tests, muscle mass and functionality as outcomes. However, a central aspect of functionality in lung cancer patients may be the muscle's ability to develop force in a short time. The present study therefore has rate of force development as a primary outcome with muscle mass and functionality as supporting outcomes. In addition, the patients in this study will perform one-leg resistance exercise with the other leg as the control leg. This will eliminate the interpersonal bias normally seen in randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* patients (men and women) from the age of 18 years and above; patients with lung cancer (NSCLC stage III - IV and SCLC ED); patients with performance stage 0-2 according to WHO criteria

Exclusion Criteria:

* Patients where the doctor has listed contraindications for physical activity in the medical record; documented bone and brain metastases; persistent medullary plasia; patients on anticoagulation treatment; diagnosed symptomatic cardiac disease, including clinical congestive heart disease, arrhythmia requiring treatment or diagnosed myocardial infarction within the last three months; pericardial exudate; patients in terminal treatment; senile dementia and psychotic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength/function: Rate of Force Development (RFD) | Baseline, 6 weeks, 12 weeks
  The between group change in Rate of Force Development (Nm/s) of the knee extensors. Assessed in the CON-TREX MJ dynamometer.

SECONDARY OUTCOMES:
Functionality: 6 minutes walk test (6-MWT) | Baseline, 6 weeks, 12 weeks
  Change in walking distance
Lean leg mass | Baseline, 6 weeks, 12 weeks
  The between group change in lean leg mass (kg) assessed by whole-body dual-energy x-ray absorptiometry (DXA) scan
Functionality: Postural balance | Baseline, 6 weeks, 12 weeks
  Postural one-leg balance on a 5-cm high, 3-cm wide, and 50-cm long plastic bar. Between group change in number of times the participants steps off the bar or needs support to prevent falling in a period of 1 min.
Functionality: Sit-to-stand (30s STS) | Baseline, 6 weeks, 12 weeks
  Change in sit-to-stand in 30 seconds
Functionality: Sit-to-stand (5reps STS) | Baseline, 6 weeks, 12 weeks
  Change in time for 5 STS repetitions
Muscle strength/function: 1 RM | Baseline, 6 weeks, 12 weeks
  The between group change in 1 repetition maximum in knee-extension and leg-press
Muscle strength/function: Power | Baseline, 6 weeks, 12 weeks
  The between group change in maximum isometric knee extension power (Nm). Assessed in the CON-TREX MJ dynamometer.
Muscle strength/function: Isokinetic strength | Baseline, 6 weeks, 12 weeks
  The between group change in maximum isokinetic knee extension power (Nm) (60 degrees/s). Assessed in the CON-TREX MJ dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Quist, ph.d., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University hospital Copenhagen, København Ø, Please Select, Denmark

IPD SHARING:
Plan to Share IPD: No